## External Fixation Versus Splinting of Acute Calcaneus Fractures

NCT04063657

May 2, 2019

# INSTRUCTIONS: use in conjunction with the online Initial Review Application form when no sponsor authored protocol is available.

## 1) Protocol Title

Title: Staged External Fixation of Acute Calcaneal Fractures

Protocol Version Date: 05/02/2019

## 2) Objectives

#### Aim:

 Determine if external fixation decreases soft tissue complications compared to splinting.

- o Determine if external fixation decreases time to definitive surgical stabilization and improves final fixation compared to splinting.
- o Determine if external fixation improves functional outcomes as evaluated by validated funcational scoring systems.

#### Hypothesis:

 External fixation improves definitive fixation and functional outcomes of acute calcaneal fractures with decreased complication rates compared to splinting

## 3) Background

Acute displaced calcaneal fractures are a regularly encountered orthopedic injury that can be complex to treat. Operative treatment of these fractures has been shown to have improved functional outcome scores compared to patients treated non-operatively.<sup>1-3</sup> Operative treatment aims to reduce the articular surface and restore radiographic parameters such as Bohler's angle, both of which have been correlated with improved long term morbidity.<sup>4-5</sup>

Within operative management options the definitive operative choice to minimize soft tissue and post-operative complications remains controversial. Minimally invasive and percutaneous fixation techniques of complex calcaneus fractures has been shown to decrease soft tissue complications compared to open reduction internal fixation (ORIF) techniques.<sup>6-7</sup> However, there is concern about the use of percutaneous techniques leading to a loss of reduction and important radiographic parameters.<sup>6</sup> Additionally, direct visualization that is offered in an open technique is often preferable.

Clinicians favoring an open technique have sought ways to minimize soft tissue complications by using a temporary external fixator as similar to the often utilized staged management of tibial plateau and tibial platfond fractures.<sup>8-10</sup> This delay is necessary for soft tissue swelling to subside prior to surgery with the external fixator allowing for prevention of early clot and fibrinous material between malaligned fracture fragments that may impede definitive reduction in the operating room. Additionally, early temporary fixation will restore native soft tissue biology and calcaneal morphology allowing for optimal healing conditions prior to definitive fixation.

Given these benefits, external fixators have been studied to treat acute calcaneus fractures definitively, in a brief-(days) or prolonged- (months) staged approach. <sup>11-15</sup> To date there has only been three case series describing a brief-staged technique with use of an external fixator for treatment of complex calcaneal fractures. <sup>16-18</sup> Our study will provide the first prospective-randomized controlled trail of this potentially practice changing protocol. The purpose of this study is to compare the efficacy of temporary external fixation vs. splinting for the treatment of acute calcaneal fractures prior to definitive surgical fixation.

#### Reference:

- 1. De boer AS, Van lieshout EM, Den hartog D, Weerts B, Verhofstad MH, Schepers T. Functional outcome and patient satisfaction after displaced intra-articular calcaneal fractures: a comparison among open, percutaneous, and nonoperative treatment. J Foot Ankle Surg. 2015;54(3):298-305.
- 2. Melcher G, Bereiter H, Leutenegger A, et al. Results of operative treatment for intra-articular fractures of the calcaneus. J Trauma 1991; 31:234–8.
- 3. Basile A. Operative versus nonoperative treatment of displaced intra- articular calcaneal fractures in elderly patients. J Foot Ankle Surg 2010;49:25–32. [55]
- 4. Loucks C, Buckley R. Bohler's angle: correlation with outcome in displaced intraarticular calcaneal fractures. J Orthop Trauma. 1999;13(8):554-8.
- 5. Waseem M. The use of subtalar arthroscopy in open reduction and internal fixation of intra-articular calcaneal fractures. Injury. 2003;34(6):475.
- 6. DeWall M, Henderson CE, McKinley TO, Phelps T, Dolan L, Marsh JL. Percutaneous reduction and fixation of displaced intra-articular calcaneus fractures. J Orthop Trauma 2010;24(8):466-72.
- 7. Jin C, Weng D, Yang W, He W, Liang W, Qian Y. Minimally invasive percutaneous osteosynthesis versus ORIF for Sanders type II and III calcaneal fractures: a prospective, randomized intervention trial. J Orthop Surg Res. 2017;12(1):10.
- 8. Sirkin M, Sanders R, DiPasquale T, Herscovici D, Jr. A staged protocol for soft tissue management in the treatment of complex pilon fractures. J Orthop Trauma 2004;18(8 Suppl):S32-8.
- 9. Thordarson DB. Complications after treatment of tibial pilon fractures: prevention and management strategies. J Am Acad Orthop Surg 2000;8(4):253-65.

- 10. Egol KA, Tejwani NC, Capla EL, Wolinsky PL, Koval KJ. Staged management of high-energy proximal tibia fractures (OTA types 41): the results of a prospective, standardized protocol. J Orthop Trauma 2005;19(7):448-55; discussion 56.
- 11. Fu TH, Liu HC, Su YS, Wang CJ. Treatment of displaced intra-articular calcaneal fractures with combined transarticular external fixation and minimal internal fixation. Foot Ankle Int 2013;34(1):91-8. [15] Begue T, Mebtouche N, Auregan JC, Saintyves G, Levante S, Cottin P, et al.
- 12. External fixation of the thalamic portion of a fractured calcaneus: a new surgical technique. Orthop Traumatol Surg Res 2014;100(4):429-32. [16] Magnan B, Bortolazzi R, Marangon A, Marino M, Dall'Oca C, Bartolozzi P.
- 13. External fixation for displaced intra-articular fractures of the calcaneum. J Bone Joint Surg Br 2006;88(11):1474-9. [17] Besch L, Waldschmidt JS, Daniels-Wredenhagen M, Varoga D, Mueller M,
- 14. Hilgert RE, et al. The treatment of intra-articular calcaneus fractures with severe soft tissue damage with a hinged external fixator or internal stabilization: long-term results. J Foot Ankle Surg 2010;49(1):8-15.
- 15. Kissel CG, Husain ZS, Cottom JM, Scott RT, Vest J. Early clinical and radio-graphic outcomes after treatment of displaced intra-articular calcaneal fractures using delta-frame external fixator construct. J Foot Ankle Surg 2011;50(2):135-40.
- 16. Githens M, Shatsky J, Agel J, Bransford RJ, Benirschke SK. Medial external fixation for staged treatment of closed calcaneus fractures: Surgical technique and case series. J Orthop Surg (Hong Kong). 2017;25(3):2309499017727915.
- 17. Farrell BM, Lin CA, Moon CN. Temporising external fixation of calcaneus fractures prior to definitive plate fixation: a case series. Injury. 2015;46 Suppl 3:S19-22.
- 18. Baumgaertel FR, Gotzen L. Two-stage operative treatment of comminuted os calcis fractures. Primary indirect reduction with medial external fixation and delayed lateral plate fixation. Clin Orthop Relat Res. 1993;(290):132-41.

### 4) Inclusion and Exclusion Criteria

#### **Inclusion Criteria Exclusion Criteria** Voluntary consent unable to consent Age 18 to 69 age < 18 Clinical and/or advanced imaging Prior surgery of the affected extremity confirming an acute calcaneal fracture that Prisoners has occurred within 2 days of which, Pregnant women eventually definitive surgery is Inflammatory arthritis recommended/accepted. Non-english speaking spatients

## 5) Study Timelines

- Study will begin after IRB approval
- Patient recruitment will take place over two years, however this may be lonher depening on the number of patients who require definitive surgery
- The duration of the subject's participation in the study will conclude at two year postoperatively
- The primarly analysis will be complete within 3 years of the study start time

## 6) Study Endpoints and Procedures involved

#### I. Design

- Subjects will be recruited from the UC Davis Medical Center. Adults diagnosed with an acute (<1-2 days from injury) calcaneal fracture recommended for operative treatment will be offered enrollment into the study.
- O A total of 100 patients will be enrolled in the study. The sample size can be calculated at 35 per treatment groups after considering multiple comparisons and using an 80% power and an  $\alpha = 0.05$ . This would require a minimum of 70 patients for the study; however, factoring in a 30% dropout rate, a minimum of 100 patients will be enrolled into the study with a minimum of 50 patients per group.

#### II. Methods

- Patients will be randomized to one of two treatment groups: temporary external fixation or temporary splinting. Both temporary treatments are those routinely used/available at the UCD health system. Subject are to wear the temporary treatment method until definitive surgery.
- Safety endpoints occur at conclusion of the definitive fixation of their calcaneal fracture.

- All subjects will receive standard perioperative and operative treatment of their injury. Patients will receive standard clinical follow up for which their healing and functional status will be continually evaluated.
- o Follow up after surgery will be at 6 time points: 2 weeks, 6 weeks, 12 weeks, 6 months, 1 year, 2 years
- The research related activities are randomization, using SOS surveys at specified time points, and collecting/reporting data regarding the outcomes from routine visits and survey responses.

#### III. Outcomes

#### **Primary outcome**

- 1. Time to definitive surgery
- 2. Soft tissue complications (at routine follow ups which are 2, 6, & 12 weeks, and 6, 12, & 24 months after surgery)

#### **Secondary outcomes**

- 1. Union rate via standard weight bearing plain radiographs (harris axial/lateral views) at 6 weeks, 12 weeks, 6 months, 1 year, and 2 years after surgery. We will also obtain a 1X CT scan of the injured foot at 1 year after surgery to monitor for arthritic progression.
- 2. Radiographic parameters(Bohler's angle, clancaneal height/width/length, and angle of Gissan)
- 3. Other complications
- 4. Clinical outcomes will be evaluated to monitor patients' activity levels, pain, and functional status. This will be done primarly using the webbased Surgical Outcome System™ (SOS)
  - The SOS is currently a UCD IRB approved study (IRB # 1192222). It is a large international web-based registry that permits collection of baseline characteristics of patients undergoing orthopedic procedures. The data is collected using direct entry into a web-based collection system called the Surgical Outcome System (SOS). By completing these surveys, the investigator surgeon has the opportunity to monitor the subjects progress after treatment, even when they are not scheduled to see the provider. The investigator surgeon will also be able compare the outcomes to the average de-identified global data.
  - In order to utilize the web-based surveys, we would invite patients to dual enroll and consent into SOS. If, the subject forgoes SOS participation, the surveys may be filled out manually and this data will not be part of SOS.
  - Subjects fill out surveys before visits at 7 total time points: preoperatively, & postoperatively at 2, 6, and 12 weeks and 6 months, 1 and 2

years. The surveys may include the Visual Analogue pain score(VAS), Patient-reported outcomes measurement information system 10 short form (PROMIS 10), or Veterans RAND 12 item Health survey (VR-12), Foot function index questionnaire (FFI-R) or Foot and Ankle Ability measure activities of daily living (FAAM ADL), and FAAM sport

- IV. **Analysis:** The data will be analyzed for differences between splinting and external fixator treatement groups. Data will be stratified and analyzed for further differences in outcomes based on other factors (ie: demographics, comorbidities..)
  - To assess significance the alpha level will be set at < 0.05.
  - Continuous data will be reported as means, standard deviation(SD), range, with 95% confidence intervals
  - Categorical data will be reported as frequencies or percentages with 95% confidence intervals

## 7) Data and/or Specimen Management and Confidentiality

☑I understand that the UC Davis Health Electronic Health Record (EMR/EPIC) also contains the clinical data for Marshall Medical Center (MMC). I understand that MMC patient data cannot be accessed for research purposes and that I must take the necessary steps to ensure that MMC data is not accessed, used, or disclosed for UC Davis Health research purposes.

Since this is a prospective study, the PI/research team are part of the data collection process. Thus, the data will be identifiable at first to the research team. However, all efforts will be made to de-identify the data. A coding system will be used to assigned a unique code to each subject. Only authorized research staff members will have access to data.

All identifiable electronic data will be maintained on an encrypted device requiring password for access. Passwords will not be shared and will be protected from access.

If protected health information or personal information from the medical records will be stored on an encrypted device, investigators will follow applicable university policies (UC Davis Hospital Policy 1313, UCDHS P&P 2300-2499, and UC Business and Finance Bulletin on Information Security (IS-3).

All paper records will be stored in a locked room/file-cabinet with access limited to only individuals who have a right and need for access.

## 8) Data and/or Specimen Banking

If the patient also provides voluntary consent to enter the SOS web-based registry, the subject will be dual consented and also enrolled into the SOS. The data will enter the main SOS global registry(de-identified).

## 9) Provisions to Monitor the Data to Ensure the Safety of Subjects

This is a minimal risk study. There are no anticipated risks specific to study participation. There are no experimental procedures and participation in this study is not anticipated to affect the medical treatment of enrolled subjects.

Subjects will be randomized into two temporary treatments are likely to benefit from either arm of the study.

Procedures performed are currently standard of clinical practice for management calcaneal fractures.

In order to protect the rights and welfare of the subjects, an initial site set-up visit will be performed to ensure proper documentation. Further monitoring (including the close out visit) will take place as needed by our internal Research staff. The PI reviews and track all complications as standard care.

## 10) Withdrawal of Subjects

- Subjects can voluntarly withdrawl at anytime
- Otherwise, the subjects are withdrawn if:
  - They have inadequate follow up without communicating with research staff.
  - o Their health changes, and staying in the study is no longer in his or her best interest
  - They do not follow the study rules or no longer meet requirments to be in the study
  - o The researchers terminate the study.

## 11) Risks to Subjects

There are no physical risks in this study.

There is the risk of randomization in this study.

There is a privacy risk, since we will record data which poses the risk of loss of confidentiality. The risk will be minimized through the processes described above. This study will abide by all applicable law, regulations, and standard

operating governing the protection of human subjects, student information and protected health information.

## 12) Potential Benefits to Subjects

These subjects are not likely to received any benefit from the proposed research, but others may benefit from the knowledge obtained

- 13) Multi-Site Research: Not applicable
- 14) Community-Based Participatory Research: Not applicable

## 15) Sharing of Results with Subjects

Subjects will be aware of the survey scores as they are self-reported. Subjects will be aware of which treatment option they receive as they are visible. The results of this study will not be shared with other subjects or others.

- 16) Prior Approvals: IRB approval
- 17) Provisions to Protect the Privacy Interests of Subjects

The subjects' privacy interests will be protected, as information will only be made available to those directly involved in the research study. The information will be stored in a password-protected spreadsheet which will have a assigned a code to protect patient confidentiality. The code will be kept separate from the data. At the completion of the data analysis, the code key will be destroyed. The subjects will feel at ease as researchers will treat them with respect and address any of their questions/concern

- **18)** Compensation for Research-Related Injury: Not applicable as study is minimal risk
- **19)** Economic Burden to Subjects: No different from routine care, and thus billed to insurance.

## 20) Drugs or Devices:

The devices used in this study is FDA approved and thus not investigational. The device will be used as intended by FDA.

## 21) Review Requirements

Are there any contractual obligations or other considerations that require IRB review of this research, or review at intervals other than those required by the Common Rule or FDA? If yes, check box: NO